CLINICAL TRIAL: NCT04866472
Title: Comparison of Video Laryngoscope (VLS) With GlideRite Ridge Stylet vs Video Laryngoscope With the TCI Articulating Indroducer for Endotracheal Intubation in Predicted Difficult Airways. A Prospective Randomized Control Trial
Brief Title: Comparison Using a VLS Using GlideRite Stylet Versus TCI Articulating Introducer in Predictive Difficult Intubation
Acronym: DA-TCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Rainer Lenhardt, Professor, University of Louisville, School of Medicine, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB20.0744
Record Dates: First submitted 2021-04-02; First posted 2021-04-29 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Predicted Difficult Airway

STUDY DESIGN:
Intervention Model Description: Randomization to Control: Video-Laryngoscope and GlideRite Rigid Stylet vs Intervention: Video-Laryngoscope with TCI Articulating Device
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Video Laryngoscope and GlideRite Ridgid Stylet (Other)
  Interventions: Device: video-laryngoscope and GlideRite Rigid Stylet
- Video Laryngoscope and TCI Articulating Introducer (Experimental)
  Interventions: Device: video-laryngoscope and TCI Articulating Introducer Device

INTERVENTIONS:
Device: video-laryngoscope and GlideRite Rigid Stylet — Once subject is in the operating room, standard monitoring will be instituted including nerve stimulator. Induction will follow standard practice.Once full muscle relaxation is confirmed with a train of four of 0/4 laryngoscopy will be preformed using a video-laryngoscope (VLS) with a #3 blade for women and a #4 blade men. Endotracheal intubation will be performed using a #7 endotracheal tube in women and # 8 in men using the GlideRite Rigid Stylet. The stylet will be shaped to the curvature of the blade of the VLS and lubricated with a water-based lubricant. After successful tracheal intubation the circuit will be connected and ventilation confirmed with capnography and auscultation.
  Arms: Video Laryngoscope and GlideRite Ridgid Stylet
Device: video-laryngoscope and TCI Articulating Introducer Device — In the operating room, standard monitoring will be instituted including nerve simulator. Induction will follow standard practice. Once full muscle relaxation is achieved (train of four of 0/4) laryngoscopy will be performed using a video-laryngoscope (VLS) using a #3 blade in women and a #4 blade in men. A #7 endotracheal tube will be used for women and a #8 for men. Endotracheal intubation will be performed by placing the tube on the back of the TCI articulating introducer, after shaft is lubricated with a water based lubricant. The tip of the TCI articulating introducer will be maneuvered into the trachea and advanced until the green zone of the introducer shaft is adjacent to the glottis. The handle of the articulating introducer will then be removed and the ETT will be advanced over the articulating introducer and into the trachea via Seldinger's technique. Once in place the respiratory circuit will be connected and confirmed with capnography and auscultation.
  Arms: Video Laryngoscope and TCI Articulating Introducer

SUMMARY:
This study will assess the feasibility of using the TCI Articulating Device with video-laryngoscope in predictive, difficult airway, endotracheal intubation cases. It is meant to show the use of this device is equivalent to using the GlideRite Rigid Stylet with video-laryngoscope.

DETAILED DESCRIPTION:
Multi-Centered, Prospective, Randomized, Control Trial

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring oral endotracheal intubation
* Age 18 years or older
* Group A Criteria (need only one of the following criteria)

  1. History of difficult intubation
  2. History of head/neck radiation and prior oral cavity, pharyngeal, or laryngeal surgery

Group B Criteria (need three or more of the following)

1. Thyromental distance <6 cm (Defined as distance measured from the thyroid notch to the tip of the jaw with the head extended and the mouth closed)
2. Sternomental distance < 12 cm (Defined as distance measured as the straight line between the upper border of the manubrium sterni and the bony point of the mentum with the head in full extension and the mouth closed
3. Oropharyngeal view: modified Mallampati scale of 3 or 4
4. Mouth opening < 4 cm
5. Protruding upper teeth (severe overbite)
6. History of radiation to the neck
7. Limited neck movement: inability to extend and flex neck >90° from full extension to full flexion or presence of cervical spine pathologies and fractures (e.g., C-collar in place)
8. Body Mass Index (BMI) >35 kg/m2
9. Neck circumference .> 40 cm in females and 43 cm in males measured at the thyroid cartilage
10. Obstructive sleep apnea diagnoses or a STOP BANG score 6 and above

Exclusion Criteria:

Any patient under the age of 18 Full stomach, Untreated hiatal hernia Uncontrolled gastroesophageal reflux disease Known tracheal narrowing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time to successful intubation using a combination of video-laryngoscope and TCI Articulating Device will be equilivant to intubation success usinging a combination of video-laryngoscope and GlideRite Rigid Stylet | time measured in seconds with an estimated time of 30 to 120 seconds from the start of intubation to endotracheal tube placement verified by CO2
  successful intubation

SECONDARY OUTCOMES:
Ease of intubation using TCI Articulating Device as compaired to GlideRite Rigid Stylet as rated by provider | completed immediately after subject intubation
  completion by provider of "Ease of Intubation" visual score scale measured from 0 to 100, with 0 being impossible intubation and 100 perfectly easy intubation
Need to use a maneuver called "corkscrew" ETT to pass glottis | Period in seconds with an estimated time of 30 to 120 seconds between start of intubation procedure to ETT placement or failure to place
  provider confirms use of "corkscrew" maneuver during or after intubation, scale as yes or no
Blood in airway | Period in seconds with an estimated time of 30 to 120 seconds between start of use of TCI Articulating Device to placement of ETT tube or failure to place
  Provider reports blood in airway after the end of the intubation
Time to intubate using either control or intervention | Time measured in seconds, with an estimated time of 30 to 120 seconds, from time of first view of glottis to time ETT placement or failure to place
  Time from first view of glottis to ETT placement or failure to place, up to three attempts using each technique

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Louisville School of Medicine, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No
Subjects will be given an identification code (study number) that will be transcribed on all subject files. A master list containing the assigned identification code and the subjects name and medical record number will be kept separately by the research coordinator. All data will be de-identified

REFERENCES:
- [Background] Mort TC. The incidence and risk factors for cardiac arrest during emergency tracheal intubation: a justification for incorporating the ASA Guidelines in the remote location. J Clin Anesth. 2004 Nov;16(7):508-16. doi: 10.1016/j.jclinane.2004.01.007. PMID 15590254
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Caplan RA, Posner KL, Ward RJ, Cheney FW. Adverse respiratory events in anesthesia: a closed claims analysis. Anesthesiology. 1990 May;72(5):828-33. doi: 10.1097/00000542-199005000-00010. PMID 2339799
- [Background] Lenhardt R, Burkhart MT, Brock GN, Kanchi-Kandadai S, Sharma R, Akca O. Is video laryngoscope-assisted flexible tracheoscope intubation feasible for patients with predicted difficult airway? A prospective, randomized clinical trial. Anesth Analg. 2014 Jun;118(6):1259-65. doi: 10.1213/ANE.0000000000000220. PMID 24842175